CLINICAL TRIAL: NCT02487693
Title: Radiofrquency Ablation Combined With Cytokine-induced Killer Cells for the Patients With Ovarian Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ovarian001
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA alone (No Intervention): Patients undergo radiofrequency ablation alone.
- RFA+CIK (Experimental): Autologous cytokine-induced killer cells were transfer via venous one week after RFA Interventions
  Interventions: Procedure: Radiofrequency ablation; Biological: Cytokine-induced killer cells

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation is performed percutaneously under CT/US guidance
  Other Names: RFA
  Arms: RFA+CIK
Biological: Cytokine-induced killer cells — The patients received autologous cytokine-induced killer cells transfusion one week after RFA treatment.
  Other Names: CIK
  Arms: RFA+CIK

SUMMARY:
The purpose of this study is to determine whether combining of radiofrequency ablation (RFA) and cytokine-induced killer cells (CIK) transfusion can prolong survival of patients with ovarian carcinoma.

DETAILED DESCRIPTION:
The primary objective is to evaluate whether RFA followed by CIK transfusion can prolong survival of patients with ovarian carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with FIGO stage II ovarian carcinoma;
2. cytoreductive surgery performed and 6 courses of platinum-based chemotherapy completed;
3. medical records maintain comprehensive data on treatment and follow-up;
4. no history of previous malignancies.

Exclusion Criteria:

1. neoadjuvant chemotherapy applied;
2. less than 6 courses of chemotherapy or more than 6 courses of chemotherapy completed;
3. medical records maintain incomplete data on treatment or follow-up;
4. history of previous malignancy.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2038-06 (Estimated); Study Completion 2040-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 1 year
  Recurrence-free survival (RFS) was defined as the time from the date of RFA to the date of recurrence or the date of the last follow-up.

SECONDARY OUTCOMES:
Adverse events | 4 weeks
  Adverse events related to RFA and CIK treatments.